CLINICAL TRIAL: NCT00160992
Title: Phase I Study of in Vivo Expansion of Melan-A/MART-1 Antigen-Specific CD8 T Lymphocytes Following Transient Immunosuppression in Patients With Advanced Melanoma
Brief Title: Adoptive Cell Transfer Combined With Peptide Vaccination in Transiently Immunosuppressed Melanoma Patients
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Fond'action contre le cancer (Unknown); Barletta Foundation (Other); NCCR (National Center of Competence in Resaerch, Switzerland) (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CePO-ITA-01
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Melanoma
Keywords: Adoptive cell transfer; peptide vaccination; melanoma; immunosuppression and homeostatic proliferation
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Biological: Melan-A analog peptide

SUMMARY:
Patients with advanced stage melanoma who underwent vaccination with the Melan-A/MART-1 peptide and who display detectable levels of Melan-A specific CD8+ T cells in peripheral blood are eligible for this trial. After collecting and freezing of these tumor specific T cells via apheresis, patients undergo a single cycle of immunosuppressive chemotherapy. 3 days after, cells are reinfused and peptide vaccination continued. The aim of this immunotherapy protocol is to boost tumor specific T cells during the immune recovery period in order to reinforce the patients' immune response against the tumor.

DETAILED DESCRIPTION:
Patients who have previously been vaccinated with Melan-A/MART-1 peptide are eligible. Whole PBMC's containing Melan-A specific CD8+ lymphocytes are collected via lymphocytapheresis and freezed. Lymphodepleting chemotherapy consists of 2 days of Busulfan 2mg/kg at days -7,-6, followed by Fludarabine 30mg/m2 at days -5,-4,-3. At day 0, whole untreated PBMC's are reinfused to the patient and vaccination with Melan-A analog peptide is restarted and repeated every 4 weeks. Immunomonitoring with detailed FACS analysis using tetramers is performed at day 0,8,15,30, and then monthly. The aim is to boost Melan-A specific CD8 T cells in vivo during homeostatic proliferation after lymphodepletion and antigen driven proliferation due to peptide vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV melanoma
* tumor expressing Melan-A
* patient of HLA-A2 subtype
* Detectable immune response after peptide vaccination with Melan-A
* Disease progression during peptide vaccination

Exclusion Criteria:

* Cerebral metastases
* rapidly progressive disease, that necessitates systemic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2004-07; Study Completion 2005-08

PRIMARY OUTCOMES:
Toxicity and feasibility

SECONDARY OUTCOMES:
Immunomonitoring of the immune reconstitution period

CONTACTS AND LOCATIONS:
Overall Officials: Verena Voelter, MD, Principal Investigator — Multidisciplinary Oncology Center, University of Lausanne Hospitals
Locations (1):
- Multidisciplinary Oncology Center, University of Lausanne Hospitals, Lausanne, Switzerland